CLINICAL TRIAL: NCT01443949
Title: Individual Differences in Reward and Impulse Control Circuitry as Risk Factors for Addiction
Brief Title: Teenagers, Drug Addiction, and Reward and Impulse Control
Status: Withdrawn | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911466; 11-DA-N466
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2013-04-04

CONDITIONS: Adolescents; Conduct Disorder; Vulnerability to Substance Addicition
Keywords: fMRI; Reward; Adolescents; Impulse Control; Cabergoline
MeSH Terms: conditions — Conduct Disorder

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background:

- The risk for becoming addicted to drugs varies from person to person, even among those who use similar drugs in a similar way. Studies suggest that certain personality traits seen in people with drug addiction may be present before drug use. These traits include responding differently to rewards or impulsivity. Early use of drugs (before age 15) is also associated strongly with drug addiction later in life. Researchers want to study teenagers with and without certain behavioral problems, including those who have used drugs and those who have not. This may help them better understand behaviors that might predict future drug addiction.

Objectives:

- To understand brain function in teenagers who may be at a higher risk than others to drug addiction.

Eligibility:

* Teenagers between 13 and 17 years of age who fit into one of four groups:
* Have never or rarely used drugs
* Have never or rarely used drugs and have conduct or behavior disorders
* Have used drugs on many occasions
* Have used drugs on many occasions and have conduct or behavior disorders

Design:

* Participants will be screened with a medical history, and physical and neurological exams. They will also have blood and urine tests. Participants will answer questions about past drug use and any current medications. They will also have a breathalyzer and carbon monoxide breath test to check for recent drug and alcohol use.
* This study requires four visits to the clinical center for magnetic resonance imaging (MRI) scans and other tests.
* The first study visit will include training for the MRI scans. Participants will practice the tasks in front of a computer and in a mock (fake) MRI machine. Participants will also be asked several questions about their personality and past experiences.
* Researchers will test changes to tryptophan and dopamine levels. Both of these chemicals affect decision making and brain function. On the three study visits, participants will have the following tests in a randomly selected order. One study will be done at each visit.
* MRI scans with changes to dopamine and tryptophan levels
* MRI scans with changes to dopamine only (with placebo)
* MRI scans with changes to tryptophan only (with placebo)
* Participants will be monitored with frequent blood draws and other tests during the study visits....

DETAILED DESCRIPTION:
Background: Even under similar drug use patterns, the risk for drug addiction varies from individual to individual. However, the neurobiological mechanisms underlying this variability are poorly understood and characterized. Studies suggest that certain traits observed in substance dependent individuals may actually precede drug use, and could augur future substance dependence. Understanding how the presence of these traits increases vulnerability to substance addiction could aid in the development of early intervention, preventative measures, as well as better treatment strategies.

Objective: The primary goal of this protocol is to improve our understanding of increased susceptibility to developing substance addiction. We focus here on reward and punishment learning, and impulse control, with an emphasis on the underlying role of dopamine and serotonin function in these two cognitive functions. Further, given that cortical plasticity is enhanced during childhood and adolescence, we begin to address whether early exposure to substances enhances neurobiological changes that make an individual vulnerable to subsequent substance addiction.

Subject Population: We focus on adolescents (13-17 years old) with known increased vulnerability to substance addiction individuals with early exposure to substances, i.e. , those who have used drugs on multiple occasions before the age of 15, and those diagnosed with conduct disorder and who are not as yet substance dependent, along with matched controls.

Experimental Design: This study involves cognitive, pharmacological and functional magnetic resonance imaging (fMRI) testing in a mixed, within/between-subject design. Based upon power analyses, we estimate needing 30 participants in each of 4 groups early exposure (EE), conduct disorder (CD-NE), conduct disorder with early exposure (CD-EE), and controls with no early exposure (NE) to complete the experiment. This is a within subjects, placebo controlled, crossover design with participants tested before and after 1) cabergoline (D2 receptor agonist) treatment, 2) acute tryptophan depletion, and 3) placebo.

Outcome Measures: The primary outcome measures will be BOLD fMRI activation and behavioral performance on various cognitive tasks that deal with impulse control and reward learning before and after each of the three treatments listed above. Secondary outcome measures include gene x environment interactions and stress and novelty-seeking measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants:

1. Between 13 and 17 years old (inclusive);
2. Must be able to provide informed assent and have a parent/guardian who can provide informed consent;
3. Blood pressure (BP) and heart rate (HR) while sitting at or below the following values after five min rest: Systolic BP (SBP) 140 mm Hg, diastolic BP (DBP) 90 mm Hg, heart rate (HR) 100 bpm;
4. 12-lead standard ECG and three-minute rhythm strip without clinically relevant abnormalities;
5. Estimated IQ (Bullet) 85 determined by the Wechsler Abbreviated Scale of Intelligence (The Psychological Corporation, 1999);
6. Right-handed (based on Edinburgh Handedness Inventory).
7. Eligible to enter the MRI scanner, as determined though self and parent (guardian) report on the MRI screening form (from the screening protocol 06-DA-N415).

Group EE:

- History of substance use on 5 or more occasions (not including over-the-counter medications and energy drinks) as assessed through the Substance Use Questionnaire.

Group CD-NE:

- History of diagnosis with conduct disorder, assessed from parental or self-report (and verified by study-clinician).

Group CD-EE:

* History of diagnosis with conduct disorder, assessed from parental or self-report (and verified by study-clinician);
* History of substance use on 5 or more occasions (not including over-the-counter medications and energy drinks) as assessed through the Substance Use Questionnaire.

EXCLUSION CRITERIA

All participants:

1. Report of a history of significant medical/neurological illness that might interfere with imaging data such as HIV positive status, cerebral vascular accident (CVA), central nervous system (CNS) tumor, traumatic brain injury, multiple sclerosis (MS) or other demyelinating diseases, epilepsy, or movement disorders;
2. History of psychosis or any current DSM-IV axis I disorder (other than simple phobia and conduct disorder);
3. Current use of psychotropic medication that may alter attentional functioning (e.g., Clonidine, antipsychotics, Venlafaxine, stimulants);
4. Current use of substances (not including over-the-counter medications and energy drinks) as assessed by self-report, carbon monoxide (CO) monitoring, alcohol breathalyzer and urine testing;
5. Pregnancy, which will be assessed by history during screening and by urine testing on scan days;
6. Claustrophobia by self and/or parent (guardian) report, or through response to the mock-scanner environment, severe enough to preclude toleration of the scanning environment.

Group NE:

* History of substance use on 5 or more occasions (not including over-the-counter medications and energy drinks) as assessed through the Substance Use Questionnaire;
* History of diagnosis with conduct disorder, assessed from parental or self-report (and verified by study-clinician).

Group EE:

- History of diagnosis with conduct disorder, assessed from parental report (and verified by study-clinician).

Group CD-NE:

- History of substance use on 5 or more occasions (not including over-the-counter medications and energy drinks) as assessed through the Substance Use Questionnaire.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-09-11; Study Completion 2013-04-04

PRIMARY OUTCOMES:
Bold fMRI activation and behavioral performance on various cognitive tasks that deal with impulse control and reward learning before and after each of the three treatments.

SECONDARY OUTCOMES:
Secondary outcome measures include gene x environment interactions and stress and novelty-seeking measures.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)

REFERENCES:
- [Background] Barr CS, Newman TK, Lindell S, Shannon C, Champoux M, Lesch KP, Suomi SJ, Goldman D, Higley JD. Interaction between serotonin transporter gene variation and rearing condition in alcohol preference and consumption in female primates. Arch Gen Psychiatry. 2004 Nov;61(11):1146-52. doi: 10.1001/archpsyc.61.11.1146. PMID 15520362
- [Background] Belin D, Mar AC, Dalley JW, Robbins TW, Everitt BJ. High impulsivity predicts the switch to compulsive cocaine-taking. Science. 2008 Jun 6;320(5881):1352-5. doi: 10.1126/science.1158136. PMID 18535246
- [Background] Belsky J, Jonassaint C, Pluess M, Stanton M, Brummett B, Williams R. Vulnerability genes or plasticity genes? Mol Psychiatry. 2009 Aug;14(8):746-54. doi: 10.1038/mp.2009.44. Epub 2009 May 19. PMID 19455150